CLINICAL TRIAL: NCT07371143
Title: Turkish Adaptation, Validity, and Reliability of the Helkimo Clinical Dysfunction Index
Brief Title: Turkish Version of Helkimo Clinical Dysfunction Index
Status: Not yet recruiting | Type: Observational
Sponsor: Sevgi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 27.03.2025/61
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Temporomandibular Disorder (TMD)
Keywords: temporomandibular disorder; helkimo clinical dysfunction Index; Turkish Adaptation, Reliability, and Validity
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Helkimo Index Study Group: Individuals who meet the inclusion criteria for the Turkish validity and reliability study of the Helkimo Clinical Dysfunction Index. All participants will undergo a comprehensive clinical examination and multiple scale assessments at baseline. To assess test-retest reliability, all participants will be re-evaluated after a two-week interval.
  Interventions: Other: Turkish Version of Helkimo Clinical Dysfunction Index and Accompanying Scales

INTERVENTIONS:
Other: Turkish Version of Helkimo Clinical Dysfunction Index and Accompanying Scales — The intervention includes a detailed clinical assessment and a series of questionnaires. Participants will provide demographic data, trauma, and surgical history. Clinical evaluation includes the measurement of pain and jaw movements. Subjective symptoms will be assessed using the Numerical Pain Rating Scale (NPRS), linear ruler, Fonseca Anamnestic Index (FAI), and Mandibular Function Impairment Questionnaire (MFIQ). The Turkish version of the Helkimo Index will be administered to test its validity and reliability. To evaluate test-retest reliability, the entire procedure will be repeated for a subgroup after 14 days.

SUMMARY:
This study aimed to translate the Helkimo Clinical Dysfunction Index (HCDI) into Turkish and to test its validity and reliability as an outcome measurement method in individuals with temporomandibular dysfunction (TMD). The study included 40 patients. Participants' pain intensity and range of jaw movement were measured, followed by the administration of the HDCI, the Fonseca Anamnestic Index (FAI), and the Mandibular Function Impairment Questionnaire (MFIQ). For test-retest reliability, the same questionnaire was administered again to the same patients two weeks later, and the FAI was used to test the validity of the questionnaire.

DETAILED DESCRIPTION:
Based on the idea of making the Helkimo Clinical Dysfunction Index (HCDI) available in Turkish, our study aimed to translate this scoring system into Turkish and to test its validity and reliability as an outcome measurement method in individuals with temporomandibular dysfunction (TMD). The study aimed to include 40 patients. Pain intensity during palpation and chewing was measured using a numerical pain rating scale (NPRS), and range of jaw movement was measured using a linear ruler. Participants were then administered the HCDI, the Fonseca Anamnestic Index (FAI), and the Mandibular Function Impairment Questionnaire (MFIQ). To assess test-retest reliability, the same questionnaire was administered again to the same patients after two weeks. The FAI was used to test the validity of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 60 years of age and having been diagnosed with TMB,
* The person must be a volunteer to participate in the study,
* The native language must be Turkish.

Exclusion Criteria:

* Having a history of malignant conditions, trauma, or surgery in the cranial and cervical region,
* Inability to cooperate,
* Regular use of analgesic and anti-inflammatory drugs,
* Having dentofacial anomalies,
* Having active inflammatory arthritis,
* Having metabolic diseases (gout, osteoporosis, Cushing's disease, and hyper/hypoparathyroidism),
* Having connective tissue, rheumatological (systemic lupus erythematosus and scleroderma), and hematological disorders (anemia and leukemia),
* Having a diagnosed psychiatric illness,
* Having received physical therapy related to TMB less than 6 months ago,
* Not being a native language of Turkish

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of individuals who visit the Umay Private Oral and Dental Health Clinic between March 2025 and May 2025. Participants will include those diagnosed with Temporomandibular Disorders (TMD) based on physical and clinical examinations by a specialist. The study will recruit adults who meet the specific inclusion criteria for the Turkish validity and reliability analysis of the Helkimo Clinical Dysfunction Index. The estimated duration of the data collection phase is 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Internal Consistency of the Turkish Helkimo Clinical Dysfunction Index | At baseline (Day 0).
  Internal consistency will be evaluated using Cronbach's alpha coefficient. A value of 0.70 or higher is considered indicative of good internal consistency for the scale and its subscales.

SECONDARY OUTCOMES:
Turkish Version of the Helkimo Clinical Dysfunction Index | Baseline (Day 0) and 14 days after the baseline assessment for test-retest reliability.
  This index is a clinical tool used to assess the severity of temporomandibular disorders (TMD) through a physical examination. It evaluates five clinical items: impaired range of mandibular mobility, impaired temporomandibular joint function, muscle pain on palpation, temporomandibular joint pain on palpation, and pain during mandibular movement. Each item is scored as 0, 1, or 5 points, with total scores ranging from 0 to 25. Higher scores indicate more severe clinical dysfunction. This measure will be used to evaluate the Turkish version's internal consistency and test-retest reliability.
Numeric Pain Rating Scale (NPRS) | Baseline (Day 0) and 14 days after the baseline assessment.
  A subjective scale where participants rate their pain during palpation and chewing from 0 (no pain) to 10 (worst possible pain).
Range of Jaw Movement | Baseline (Day 0) and 14 days after the baseline assessment.
  The range of jaw movement, including maximum mouth opening, protrusion, and lateral excursions, will be measured in millimeters (mm) using a linear ruler. These measurements are used to determine the mobility sub-score of the Helkimo Clinical Dysfunction Index.
Mandibular Function Impairment Questionnaire (MFIQ) Score | Baseline (Day 0) and 14 days after the baseline assessment.
  A questionnaire consisting of 17 items to evaluate functional limitations in mandibular movements (e.g., chewing, speaking, yawning). Each item is scored from 0 (no difficulty) to 4 (impossible to perform). Higher total scores indicate a greater level of functional impairment.
Fonseca Anamnestic Index (FAI) Score | Baseline (Day 0) and 14 days after the baseline assessment.
  A multidimensional tool consisting of 10 items used to assess jaw function limitations, pain frequency, and parafunctional behaviors related to TMD. Each item is answered as "yes" (10 points), "no" (0 points), or "sometimes" (5 points). Total scores range from 0 to 100, where higher scores indicate greater severity of TMD. Severity is classified as: 0-15 (no TMD), 20-40 (mild), 45-65 (moderate), and 70-100 (severe TMD). This index will be used to evaluate concurrent validity with the Helkimo Index.

CONTACTS AND LOCATIONS:
Locations (1):
- Umay Private Oral and Dental Health Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yildiz NT, Alkan A, Kulunkoglu BA. Validity and Reliability of the Turkish Version of Mandibular Function Impairment Questionnaire. Cranio. 2024 Mar;42(2):160-170. doi: 10.1080/08869634.2021.2004715. Epub 2021 Nov 18. PMID 34789075
- [Result] Stegenga B, de Bont LG, de Leeuw R, Boering G. Assessment of mandibular function impairment associated with temporomandibular joint osteoarthrosis and internal derangement. J Orofac Pain. 1993 Spring;7(2):183-95. PMID 8358365
- [Result] Kaynak BA, Tas S, Salkin Y. The accuracy and reliability of the Turkish version of the Fonseca anamnestic index in temporomandibular disorders. Cranio. 2023 Jan;41(1):78-83. doi: 10.1080/08869634.2020.1812808. Epub 2020 Aug 25. PMID 32840464
- [Result] Bevilaqua-Grossi D, Chaves TC, de Oliveira AS, Monteiro-Pedro V. Anamnestic index severity and signs and symptoms of TMD. Cranio. 2006 Apr;24(2):112-8. doi: 10.1179/crn.2006.018. PMID 16711273
- [Result] van der Weele LT, Dibbets JM. Helkimo's index: a scale or just a set of symptoms? J Oral Rehabil. 1987 May;14(3):229-37. doi: 10.1111/j.1365-2842.1987.tb00714.x. PMID 3474383
- [Result] Alonso-Royo R, Sanchez-Torrelo CM, Ibanez-Vera AJ, Zagalaz-Anula N, Castellote-Caballero Y, Obrero-Gaitan E, Rodriguez-Almagro D, Lomas-Vega R. Validity and Reliability of the Helkimo Clinical Dysfunction Index for the Diagnosis of Temporomandibular Disorders. Diagnostics (Basel). 2021 Mar 8;11(3):472. doi: 10.3390/diagnostics11030472. PMID 33800185
- [Result] Çınar, F., Şengül, H., Çapar, H., Çakmak, C., & Bilge, Y. (2018). Perception of health news: a scale development study. J Acad Res Nurs, 4(3), 164-171.
- [Result] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561